CLINICAL TRIAL: NCT00014742
Title: Phase III Randomized Study of Collagenase in Patients With Residual Stage Dupuytren's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: State University of New York (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/15764; SUNY-SB-FDR001437
Record Dates: First submitted 2001-04-10; First posted 2001-04-11 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-04

CONDITIONS: Dupuytren's Contracture
Keywords: Dupuytren's disease; arthritis & connective tissue diseases; rare disease
MeSH Terms: conditions — Dupuytren Contracture; Arthritis; Connective Tissue Diseases; Rare Diseases | interventions — Collagenases

INTERVENTIONS:
Drug: collagenase

SUMMARY:
OBJECTIVES: I. Compare the safety and efficacy of clostridial collagenase vs placebo in terms of improving the degree of flexion deformity, range of finger motion, and grip strength in patients with residual stage Dupuytren's disease.

II. Compare the overall clinical success rate, time to return to normal finger contracture to within 0-5 degrees of normal (zero degrees), and frequency of cord rupture in the joint of patients treated with these regimens.

III. Compare the baseline change in degree of finger flexion deformity, range of motion of the treated finger, and strength of hand grip (in pounds) in patients treated with these regimens.

IV. Compare the frequency distribution of the number of patients with reduction in finger contracture to within 0-5 degrees of normal (zero degrees) and the number who require re-treatment with open-label collagenase after treatment with these regimens.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, investigator-blinded, placebo-controlled, multicenter study. Patients are randomized to one of two treatment arms.

Arm I: Patients receive a single collagenase injection into the target finger cord on day 0.

Arm II: Patients receive a single placebo injection as in arm I.

Both arms: After the 1 month evaluation, patients who are unresponsive to treatment may receive monthly injections of collagenase for a maximum of 5 injections.

Beginning at 1 day after completion of treatment, patients use a joint nighttime extension splint for 4 months and perform finger flexion/extension exercises.

Patients are followed at 1, 7, and 14 days, monthly for 3 months, every 3 months for 9 months, and then annually for 4 years.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of residual stage Dupuytren's disease with fixed flexion deformity of the finger(s) of at least 20-30 degrees caused by a palpable cord

Positive table-top test (inability to simultaneously place affected finger and palm flat against a table top)

--Prior/Concurrent Therapy--

At least 30 days since prior surgery for Dupuytren's disease At least 30 days since prior participation in a trial with an investigational drug

--Patient Characteristics--

Hematopoietic: No history of hematologic disease

Hepatic: No history of hepatic disease

Renal: No history of renal disease

Cardiovascular: No congestive heart failure, angina, or myocardial infarction within the past 6 months

Pulmonary: No history of respiratory disease

Other:

* Not immunocompromised
* HIV negative
* No history of significant illness (e.g., endocrine or neurologic disease)
* No psychosis
* No history of illicit drug abuse or alcoholism within the past year
* No infectious illness within the past 2 weeks
* No chronic or debilitating disease
* No IgE antibodies to collagenase exceeding 15 ng/mL
* No known allergy to collagenase or any of the inactive ingredients in the drug
* No other condition or circumstance that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Study Completion 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence C. Hurst, Study Chair — State University of New York